CLINICAL TRIAL: NCT00597740
Title: Clinical Utility of Propofol Sedations Without and With a Formal "ICU Sedation Protocol" in Intubated Neurotrauma Patients
Brief Title: Propofol Sedation Study
Acronym: SPIN
Status: Completed | Type: Observational
Sponsor: Scottsdale Healthcare (Other)
Responsible Party: Principal Investigator, Steven Logan, Research Compliance Administrator, Scottsdale Healthcare
Other Study IDs: 2007-106
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of Protocol: The purpose of this study will be to compare the clinical utility of Propofol sedation with and without the use of the ICU Sedation Protocol. Patients will be treated according to the attending/consulting preference. No attempt will be made to influence the patient's routine care and management. The study will compare the average hourly infusion rates for the Propofol administration, as well as obtain the nursing staffs evaluation regarding the ease of neurological assessment during each 12 hour shift

DETAILED DESCRIPTION:
Study Objectives and Design: Propofol is a short-acting sedative that is easily titratable, and is approved for use in ventilated patients. The clinical usefulness of continuous intravenous infusion of Propofol has been demonstrated in the management of ventilated ICU patients. In addition, its short duration of action permits repeated neurological assessments to be carried out in patients with neurotrauma.

Despite these benefits, Propofol is not without some drawbacks, including a lack of analgesic effects, dose dependent lowering of blood pressure, and significant expense. To address these issues, the PI developed an ICU Sedation Protocol that combines a titrated continuous infusion of intravenous morphine sulfate with the Propofol infusion to achieve the desired level of sedation. This ICU Sedation Protocol has been approved for use at Scottsdale Healthcare since 2004, and printed copies are available at all ICU nursing stations on the Osborn campus.

At the present time, the ICU Sedation Protocol is used regularly by only two of the five neurosurgeons that care for the neurotrauma patients at the Osborn campus. The remaining three neurosurgeons prefer to use a continuous Propofol infusion with intermittent doses of intravenous morphine sulfate.

The purpose of the study will be to compare the clinical utility of Propofol sedation with and without the use of the ICU Sedation Protocol. Patients will be treated according to the attending neurosurgeons preference. No attempt will be made to influence the patient's routine care and management. The study will compare the average hourly infusion rates for Propofol administration, as well as evaluating the difficulty of neurological assessment, and the ease of weaning to extubation.

This is a prospective, non-randomized, open treatment protocol open to ICU patients at Scottsdale Healthcare Osborn. Only patients with neurotrauma that require intubation will be eligible for enrollment. Patients will be treated according to the consulting neurosurgeons preference. No attempt will be made to influence the patient's routine care and management, as already stated. The choice of sedation type and use of the ICU Sedation Protocol will be at the consulting neurosurgeons discretion.

Involvement in the protocol will cease when continuous intravenous sedation is discontinued for more than 24 hours, the patient is extubated or undergoes tracheostomy, or is transferred from the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 (inclusive)
* Admitted to trauma service
* Intubated and on respiratory support
* Neurosurgical consultation for closed head injury and/or spinal trauma
* Informed consent from next of kin or POA

Exclusion Criteria:

* Patients less than 18 or more than 80 years of age
* GCS of 3 with bilaterally fixed and dilated pupils
* Penetrating head trauma (e.g., gun shot wounds, nail gun injuries, etc.)
* Pregnant women
* Mentally impaired.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurotrauma ICU patients brought to our level one trauma facility requiring intubation.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zabramski, MD, Principal Investigator — Scottsdale Healthcare Osborn - Neurosurgery
Locations (1):
- Scottsdale Healthcare Osborn, Scottsdale, Arizona, United States